CLINICAL TRIAL: NCT03697161
Title: A Phase 2, Randomized, Double-Blind, Parallel-Group Study Evaluating the Safety, Tolerability, and Efficacy of OV101 in Fragile X Syndrome
Brief Title: A Study of OV101 in Individuals With Fragile X Syndrome
Acronym: ROCKET
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Healx AI (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OV101-17-001
Record Dates: First submitted 2018-10-01; First posted 2018-10-05 (Actual); Results first posted 2024-01-23 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2023-12

CONDITIONS: Fragile X Syndrome (FXS)
MeSH Terms: conditions — Fragile X Syndrome | interventions — gaboxadol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- OV101 (gaboxadol) Regimen 1 (Experimental): Once Daily
  Interventions: Drug: OV101 (gaboxadol)
- OV101 (gaboxadol) Regimen 2 (Experimental): Twice Daily
  Interventions: Drug: OV101 (gaboxadol)
- OV101 (gaboxadol) Regimen 3 (Experimental): Three Times Daily
  Interventions: Drug: OV101 (gaboxadol)

INTERVENTIONS:
Drug: OV101 (gaboxadol) — OV101 (gaboxadol)

SUMMARY:
The purpose of this study is to assess the safety, tolerability and efficacy of oral OV101 (gaboxadol) in subjects with Fragile X syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Is male and 13 to 22 years old (inclusive) at the time of informed consent.
* Has a diagnosis of FXS with a confirmed FMR1 full mutation (≥200 CGG repeats).

Exclusion Criteria:

* Concomitant disease or condition that are clinically significant and would limit study participation
* Clinically significant lab abnormalities or vital signs at the time of screening
* History of uncontrollable seizure disorder or seizure episodes within 6 months of screening or change in the anticonvulsant pharmacotherapy in the past 3 months.
* Unable or does not have a caregiver able to comply with study requirements.
* Enrolled in any clinical trial within the 30 days before screening.

Ages: 13 Years to 22 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 36 (Actual)
Dates: Start 2018-09-17 (Actual); Primary Completion 2020-02-03 (Actual); Study Completion 2020-02-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amit Rakhit, MD, Study Director — Healx AI
Locations (6):
- United States (6):
  - Ovid Therapeutics Investigative Site, Sacramento, California
  - Ovid Therapeutics Investigative Site, Aurora, Colorado
  - Ovid Therapeutics Investigative Site, Chicago, Illinois
  - Ovid Therapeutics Investigative Site, Baltimore, Maryland
  - Ovid Therapeutics Investigative Site, Cincinnati, Ohio
  - Ovid Therapeutics Investigative Site, Nashville, Tennessee

REFERENCES:
- [Derived] Budimirovic DB, Dominick KC, Gabis LV, Adams M, Adera M, Huang L, Ventola P, Tartaglia NR, Berry-Kravis E. Gaboxadol in Fragile X Syndrome: A 12-Week Randomized, Double-Blind, Parallel-Group, Phase 2a Study. Front Pharmacol. 2021 Oct 8;12:757825. doi: 10.3389/fphar.2021.757825. eCollection 2021. PMID 34690787

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled in 7 study centers in the United States and 1 study center in Israel.
Groups:
- OV101 (Gaboxadol) Regimen 1: 5 mg/day (5 mg QD) OV101 (gaboxadol)
- OV101 (Gaboxadol) Regimen 2: 10 mg/day (5 mg BID) OV101 (gaboxadol)
- OV101 (Gaboxadol) Regimen 3: 15 mg/day (5 mg TID) OV101 (gaboxadol)
Period: Overall Study
Arm/Group | OV101 (Gaboxadol) Regimen 1 | OV101 (Gaboxadol) Regimen 2 | OV101 (Gaboxadol) Regimen 3
Started | 7 | 8 | 8
Completed | 6 | 7 | 7
Not Completed | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | OV101 (Gaboxadol) Regimen 1 | OV101 (Gaboxadol) Regimen 2 | OV101 (Gaboxadol) Regimen 3 | Total
Number analyzed (Participants) | 7 | 8 | 8 | 23
Age, Customized [Count of Participants; unit: Participants] — Population: 23 Participants
  Participants
    Age of subjects: Adolescent (13 to 17) | 4 | 5 | 4 | 13
    Age of subjects: Adult (18 to 23) | 3 | 3 | 4 | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 7 | 8 | 8 | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Black or African American | 0 | 1 | 0 | 1
  White | 7 | 7 | 6 | 20
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 3 | 8 | 8 | 19
  Israel | 4 | 0 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAE)
Description: Number of Participants with Treatment Emergent Adverse Events
Time Frame: Week 12
Measure: Number; unit: participants
Groups:
- OV101 (Gaboxadol) (5 mg QD): 5 mg/day (5 mg QD) OV101 (gaboxadol)
- OV101 (Gaboxadol) (5 mg BID): 10 mg/day (5 mg BID) OV101 (gaboxadol)
- OV101 (Gaboxadol) (5 mg TID): 15 mg/day (5 mg TID) OV101 (gaboxadol)
Arm/Group | OV101 (Gaboxadol) (5 mg QD) | OV101 (Gaboxadol) (5 mg BID) | OV101 (Gaboxadol) (5 mg TID)
Number analyzed (Participants) | 7 | 8 | 8
participants
  Any serious TEAE | 0 | 0 | 0
  Any study medication-related TEAE | 1 | 5 | 2
  Any study medication-related serious TEAE | 0 | 0 | 0
  Severity of TEAE Mild | 1 | 6 | 6
  Severity of TEAE Moderate | 0 | 2 | 0
  Severity of TEAE Severe | 0 | 0 | 0
  Any TEAE leading to discontinuation | 0 | 1 | 0
  Any TEAE leading to dose modification | 0 | 1 | 0
  Any TEAE with outcome of death | 0 | 0 | 0

2. Other Pre Specified Outcome: Clinical Global Impressions- Improvement (CGI-I)
Time Frame: Week 12
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: All adverse events collected as part of the study are reported in the Adverse Event module
Groups:
- OV101 (5 mg QD): mg/day (5 mg QD) OV101
- OV101 (5 mg BID): 10 mg/day (5 mg BID) OV101
- OV101 (5 mg TID): 15 mg/day (5 mg TID) OV101
Arm/Group | OV101 (5 mg QD) | OV101 (5 mg BID) | OV101 (5 mg TID)
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 1/7 | 8/8 | 8/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OV101 (5 mg QD) (N=7) | OV101 (5 mg BID) (N=8) | OV101 (5 mg TID) (N=8)
NASOPHARYNGITIS (Infections and infestations) | 0 (0) | 1 (4) | 1 (6)
IRRITABILITY (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
DIARRHOEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 3 (3) | 1 (1)
STEREOTYPY (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
FOOD POISONING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
VOMITING (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
VIRAL RHINITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
AGGRESSION (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
COMPULSIONS (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
DIZZINESS (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
HEADACHE (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
FEELING ABNORMAL (General disorders) | 0 (0) | 0 (0) | 1 (1)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
RASH (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-03-27): https://cdn.clinicaltrials.gov/large-docs/61/NCT03697161/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-06): https://cdn.clinicaltrials.gov/large-docs/61/NCT03697161/SAP_001.pdf